CLINICAL TRIAL: NCT05945069
Title: Feasibility of Dynamic Muscle Stimulation (DMSt) Combined with Radiofrequency (RF) for Improving Blink Quality in Subjects with Dry Eye Disease (DED)
Brief Title: Feasibility of Dynamic Muscle Stimulation + Radiofrequency for Improving Blink Quality in Subjects with Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-VBU-TRILIFT-23-01
Record Dates: First submitted 2023-06-22; First posted 2023-07-14 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Eyelid Diseases; Eyelid Movement Disorders; Dry Eye; Dry Eye Syndromes; Skin Laxity
MeSH Terms: conditions — Eyelid Diseases; Dry Eye Syndromes; Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TriLift (Experimental): Combination of Dynamic Muscle Stimulation and Radiofrequency
  Interventions: Device: TriLift device

INTERVENTIONS:
Device: TriLift device — Dynamic Muscle Stimulation combined with tripolar Radiofrequency, administered on the skin of the inferior orbital rim and below the lower eyelids

SUMMARY:
To demonstrate that DMSt + RF improves eye blink quality in subjects with dry eye disease

DETAILED DESCRIPTION:
The purpose of the study is to demonstrate that a combination of DMSt and RF applied on the periocular skin below the lower eyelids improves eye blink quality in subjects with moderate to severe signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to read, understand and sign an Informed Consent Form (ICF)
* 22 or older
* Lower lid laxity, as clinically judged with lower lid DT and the snapback test
* Moderate to severe OSDI (larger or equal to 23)
* TBUT smaller or equal to 5 sec in both eyes

Exclusion Criteria:

* Abnormally high blink rate, as estimated by the study investigator
* Any ocular surgery or eyelid surgery, within 3 months prior to screening
* Blepharoptosis
* Moderate or Severe Floppy Lid Syndrome
* Corneal Dystrophy
* Exophthalmos
* Thyroid Eye Disease
* Ocular Chemical Injury or burn
* Limbal Stem Cell Deficiency
* Facial Nerve Palsy
* Blepharospasm
* Hemifacial Spasm
* Corneal neuropathy
* Pregnant or nursing women
* Participation in a different study
* Any condition revealed whereby the study investigator deems the subject inappropriate for this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Impaired blink quality | 7 weeks after baseline (4 weeks after the 4th treatment)
  binary (yes/no) variable, based on clinical estimation of the study investigator who will use a combination of two complementary tests (the lower lid distraction test and the snap-back test) to reach a yes/no decision.

OTHER OUTCOMES:
Eyelid appearance | 7 weeks after baseline (4 weeks after the 4th treatment)
  Biomicroscopy with the slit lamp; normal, mild, moderate, severe
Overall blink quality | 7 weeks after baseline (4 weeks after the 4th treatment)
  Subjectively assessed by the study investigator; normal, mildly impaired, moderately impaired, severely impaired
Margin to Reflex Distances MRD1 and MRD2 | 7 weeks after baseline (4 weeks after the 4th treatment)
  Distances from the margins of the upper and lower lids to the central corneal reflex, in millimeters
modified Meibomian Gland Score | 7 weeks after baseline (4 weeks after the 4th treatment)
  15 meibomian glands along the lower lid (5 nasal + 5 central + 5 temporal) will be gently expressed with the dedicated expression forceps. Each gland will be scored 0 to 3, as follows: 0 = clear liquid meibum; 1 = cloudy liquid meibum; 2 = inspissated meibum; 3 = blocked). The modified Meibomian Gland score will be evaluated as the sum of scores for these 15 glands. Hence, the minimal value is 0 (all 15 glands express a clear liquid meibum), and the maximal value is 45 (all 15 glands are blocked). A decrease in the modiified Meibomian Gland Score means that the functionality of meibomian glands improved, and that the condition of the patient improved.
Ocular Surface Disease Index | 7 weeks after baseline (4 weeks after the 4th treatment)
  Symptoms will be self-evaluated with the Ocular Surface Disease Index questionnaire. Twelve (12) questions will be asked about visual difficulties experienced by the subject during the past week. Each question will be scored 0 (none of the time), 1 (some of the time), 2 (half of the time), 3 (most of the time) or 4 (all the time). The Ocular Surface Disease Index will be calculated as the sum of scores times 25, divided by the number of questions answered. An increase in the Ocular Surface Disease Index means that the symptoms are reduced and that the condition of the patient improved.
Corneal sensitivity | 7 weeks after baseline (4 weeks after the 4th treatment)
  Measured with an esthesiometer; device settings: 1 to 6
Blink rate | 7 weeks after baseline (4 weeks after the 4th treatment)
  Blinks per minute during a video-watching task
Degree of eyelid closure | 7 weeks after baseline (4 weeks after the 4th treatment)
  full, or maximal vertical height of the palpebral fissure measured in mm
Teat Breakup time | 7 weeks after baseline (4 weeks after the 4th treatment)
  Time between full blink and first appearance of a break in a fluorescein-stained eye
Adverse events | Throughout the study and up to 7 weeks after baseline (4 weeks after the 4th treatment)
  Incidence and type of adverse events
BCVA | At baseline, at 1 week after baseline (immediately before the second treatment), at 2 weeks after baseline (immediately before the third treatment), at 3 weeks after baseline (immediately before the fourth treatment) and at 7 weeks after baseline
  Best-corrected visual acuity, using an ETDRS chart (20/20, 20/25, 20/32,20/40,20/50,20/63, 20/80, 20/100, 20/200, 20/400, where 20/20 is considered perfect vision and 20/400 is considered legal blindness)
Pain/Discomfort | Immediately after a treatment session
  Pain.discomfort will be self-reported with a visual analog scale (0 to 100), with 0 representing no pain/discomfort and 100 representing intolerable pain/discomfort. A decrease in this visual analog score represents an improvement in the perception of pain/discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: James G Chelnis, MD, Principal Investigator — Manhattan Face and Eye
Locations (1):
- Manhattan Face and Eye Cosmetic and Orbital Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No